CLINICAL TRIAL: NCT07170553
Title: Digital Game Intervention for Relationship Enhancement Among Parent Child Dyads
Brief Title: Relationship Enhancement Digital Game
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Anna Queiroz, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20250185
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Parent-Child Relations; Parenting; Attachment Disorder
Keywords: Digital Intervention; Attachment Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caregiver Child Digital Intervention Group (Experimental): Participants in this group will engage with the intervention for up to 1 hour.
  Interventions: Behavioral: Digital Game
- Control Group (Active Comparator): Participants in this group will receive information about play based attachment activities and participate for up to 1 hour.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Digital Game — Parent-child dyads will come to the research site once and participate for up to one hour. Dyads will engage with a digital game prototype. The game involves brief relationship enhancing activities focused on different domains of attachment with the purpose of facilitating appropriate and healthy playful interaction between parents and children.
  Arms: Caregiver Child Digital Intervention Group
Behavioral: Control — Parent-child dyads will come to the research site once and participate for up to one hour. Dyads will receive pamphlets with information regarding play based attachment activities and be given the chance to engage in said activities.
  Arms: Control Group

SUMMARY:
The purpose of this study is to test a new digital game. Specifically, this study will aim to evaluate a digital game prototype designed to facilitate playful interactions between parents and children. The prototype will incorporate activities grounded in relationship enhancement principles. Additionally, this study will check how well using digital tools helps build strong connections, makes people get along better, and boosts parents' confidence and parenting skills.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver-child dyads.

Exclusion Criteria:

* Participant is not part of a caregiver- child dyad.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-05 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Parental Self-Efficacy as Measured by TOPSE | Baseline, Up to 1.5 hours (immediately after intervention).
  Tool to Measure Parenting Self-Efficacy (TOPSE) Total scores range from 0-480 for the complete measure. Higher scores indicate greater levels of perceived parental self-efficacy.

SECONDARY OUTCOMES:
Perceived Closeness in the Parent-Child Relationship as measured by the Social Connectedness Scale | Baseline, Up to 1.5 hours (immediately after intervention).
  Social Connectedness Scale scores range from 9 - 54. Higher scores represent greater perceived connectedness.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Queiroz, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No